CLINICAL TRIAL: NCT02743208
Title: Evaluation of a Short Femoral Stem in Total Hip Arthroplasty. A Comparative Study on Stability, Bone Remodelling and Patient Outcome.
Brief Title: Evaluation of a Short Femoral Stem in Total Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: problem due to new regulations for CE-marking of implants; lack of funding
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/846
Record Dates: First submitted 2016-03-31; First posted 2016-04-19 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty, Replacement, Hip; Surgical Procedures, Operative; Hip Prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furlong Evolution femoral stem (Experimental): Short stem hip arthroplasty (SHA) using a Furlong Evolution femoral stem, and a Furlong H-A.C. Cortical Scree Fit (CSF) plus acetabular cup system.
  Interventions: Device: Short stem hip arthroplasty (SHA)
- Furlong H-A.C. femoral stem (Active Comparator): Total hip arthroplasty (THA) using a Furlong H-A.C. femoral stem, and a Furlong H-A.C. CSF plus acetabular cup system.
  Interventions: Device: Total hip arthroplasty (THA)

INTERVENTIONS:
Device: Short stem hip arthroplasty (SHA) — Furlong Evolution femoral stem
  Arms: Furlong Evolution femoral stem
Device: Total hip arthroplasty (THA) — Furlong H-A.C. femoral stem
  Arms: Furlong H-A.C. femoral stem

SUMMARY:
In recent years, short femoral stems have been introduced. Short stems are designed based on traditional stems with good clinical results. The assumed benefit of short stems is that they are easier to use in mini-invasive surgery, and that preservation of proximal periprosthetic bone stock is better. Preservation of periprosthetic bone in the proximal femur is thought to secure long time anchoring of the implant, and reduce the risk of loosening. In addition, a good proximal bone stock makes later revision surgery less technically demanding. However, the short stem design could compromise the stability of the prosthesis, and there has been reported diverging results regarding correct positioning of short stems. This may be due to the lack of inherent aiming provided by the tip of the traditional long stems. We want to clinically evaluate the stability and bone remodelling pattern of a new short femoral stem based on a standard stem with excellent long time results. In addition we will compare the two different stems regarding positioning, when using a newly developed guiding broach for the short stem, and the standard broach for the long stem. Finally, patient reported clinical outcome scores will be evaluated with respect to implant and biomechanical reconstruction.

The aim of this study is to evaluate whether this specific short femoral stem is stable, safe to use, and if it provides the expected beneficial effects on bone remodelling.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a successful treatment of osteoarthritis and other destructive diseases of the hip joint, relieving pain and restoring the function of the joint. In Norway more than 7000 patients undergo primary hip replacement every year, and the incidence is increasing.

The femoral component of a hip prosthesis is traditionally anchored to the femoral bone with a stem introduced into the femoral canal and fixated with cement, or through bony ingrowth. Over the recent years, short femoral stems have been introduced, among other reasons to meet the increasing popularity of mini-invasive surgical procedures. The short stems are meant to be easier to introduce through a small incision like used in muscle conserving anterior and posterior approaches. Secondly, and biomechanically relevant, an important design related benefit of the short femoral stems is thought to prevent periprosthetic bone resorption. Bone remodels as a response to mechanical loading. When a stiff implant is inserted into the femoral canal, the load will "bypass" the proximal femur through the implant, and is transferred to bone distally. This results in a negative bone remodelling in the proximal femur, which leads to bone resorption, often termed as "stress shielding". Stress shielding is observed around most uncemented implants, and mainly occurs within the first 6 - 24 months postoperatively. The extent of implant coating, the material stiffness, design and the size of the stem are found to influence the degree of stress shielding. The short stems are thus designed based on the theory that proximal load transfer preserves metaphyseal bone.

Loss of proximal bone stock due to stress shielding is a controversial subject, but has several possible consequences. The exact clinical implications are not entirely determined, but periprosthetic fractures and more challenging revision surgery are recognized problems. In a revision setting it is favourable to have good proximal bone stock to achieve primary stability of the implant. Peroperative fracture and compromised stability of the implant may be a potential problem in stress-shielded bone. Furthermore, already stress-shielded bone in the proximal femur may give wear debris easier access to the interface between implant and bone, resulting in further osteolysis. Short-term results for short-stemmed implants are encouraging in some clinical papers, but most of the available implants lack long-time clinical documentation. Most papers on stress shielding are not randomized trials between long and short stems. There are a few reports of increased revision rate and challenging surgical procedures.

Uncemented prosthetic hip implants are dependent on excellent primary stability to achieve osseointegration and long-term stability. It is recognized that excessive micromotion at the bone-implant interface is associated with formation of a soft tissue and loosening of implants. Micromotion above 40μm leads to partial bone ingrowth, while values above 150μm completely inhibit bone ingrowth. The main concern in short femoral stems is that stability might be compromised. This might be due to the relatively less contact surface. There are no long term results on stability of short femoral stems available, but in vitro studies shows no significant reduction in stability of prostheses with comparable stem length to the Furlong Evolution.

Malpositioning may result in a discrepancy between the reconstructed and the native biomechanical anatomy of the hip. Altered biomechanical properties may influence the clinical outcome and survival of implants. It has been shown that horizontal femoral offset, increases significantly more using a short femoral stem compared to conventional femoral stems. Compared to the contralateral hip, horizontal femoral offset was significantly increased only when using short stems. Increased femoral offset increases the torsion forces along the stem, which in turn raises the need for primary stability to avoid micromotion. It is also shown that a short stem has a wider range of varus-valgus in the stem-shaft axis, On the other there were found no significant differences in biomechanical reconstruction of the hip when using a "broach only" short stem, or a "ream and broach" standard stem.

If there are significant differences in the biomechanical hip reconstruction, will this affect patient reported outcome?

ELIGIBILITY:
Inclusion Criteria:

* receiving primary total hip arthroplasty due to osteoarthritis, posttraumatic arthritis, avascular necrosis, or developmental hip dysplasia (Crowe grade 1)

Exclusion Criteria:

* osteoporosis
* pregnancy
* musculoskeletal problems compromising rehabilitation
* corticosteroid treatment
* dementia
* developmental dysplasia (Crowe grade II-IV)
* osteosynthesis in place
* revision surgery
* joint infection
* malignancy of the femur/pelvis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in periprosthetic bone mineral density (BMD) | 2 years
  Postoperative change in BMD following bone remodelling measured by dual-energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Migration of femoral stem | 2 years
  Migration of femoral stem measured by radiostereometric analysis (RSA)
Biomechanical reconstruction of hip anatomy | 2 years
  Biomechanical key measures in hip anatomy after reconstruction of the hip joint, compared to native anatomy in contralateral hip is analysed on a metric scale to compare the following positions: Horizontal centre of rotation. Vertical centre of rotation. Horizontal femoral offset. Vertical femoral offset. Abductor lever arm. Limb length. Stem-shaft angle, or valgus/varus.
Hip disability osteoarthritis outcome score (HOOS) | 2 years
Harris hip score | 2 years
Health-related quality of life (EQ-5D). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olav Foss, md phd, Study Director — St. Olavs Hospital

IPD SHARING:
Plan to Share IPD: No